CLINICAL TRIAL: NCT04630587
Title: Longevity of Dental Fillings by Chairside Technique Utilizing 3D Printing vs. Direct Composite Fillings
Brief Title: Longevity of Dental Fillings Utilizing 3D Printing
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: University of Helsinki (Other); Oulu University Hospital (Other); University of Turku (Other); University of Eastern Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2924410-5
Record Dates: First submitted 2020-10-26; First posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Dental Restoration Failure of Marginal Integrity; Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Each patient requires pairwise number of restorations. The randomizations are performed by each tooth to be restored by direct technique vs. indirect technique utilizing 3D printing.
Who Masked: Outcomes Assessor
Masking Description: Restorations are rated independently by blinded dentists who are not involved with the insertion of the indirect and the direct restorations and are unaware of the group status of the fillings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indirect restorations (Experimental): For the indirect technique, the cavities are prepared according to the common principles for inlays/onlays. Digital impressions are taken of each tooth with a digital impression system (3Shape TRIOS® Intraoral Scanner).The dentist, utilizing the scanner's CAD SW, designs the 3D restoration. The design is imported from the scanner SW into the Rayo 3DToothFill SW to manufacture the mould and the restoration. After printing the mould, it is transferred to the Rayo robot which manufactures the restoration by casting filling material layers in the mould. The automated filling and curing procedures in the Rayo 3DToothFill robot are directed by Rayo 3DToothFill SW. After the manufacturing process is finished, the dentist cements the finished restoration into the cavity with a dual-cure resin cement (G-CEM LinkAce®).The indirect fillings are manufactured chair-side from the same composite material as in the direct technique.
  Interventions: Procedure: Indirect restorations
- Direct restorations (Active Comparator): The direct composite restorations are performed based on normal treatment practices. For both direct and indirect restorations, commercially available short-fibre reinforced composite material (everX Flow, GC) is used for core material (replacing dentin) and flowable composite material (G-ænial® Universal Injectable, GC) for surface (replacing enamel), according the manufacturer´s instructions. The occlusion and articulation are checked and adjusted, and the restoration is finished with polishing instruments.
  Interventions: Procedure: Indirect restorations

INTERVENTIONS:
Procedure: Indirect restorations — see the Arm description

SUMMARY:
The aim of the present study is to compare the success of dental fillings prepared using 3D printing technique to those manufactured with the direct composite technique. A total of 100 adult patients will be selected from dental patients attending Kaarina Municipal Health Care Centre from October 2020. The inclusion criteria are as follows: presence of multiple cavities, fractures or cosmetic demands on bilateral permanent teeth. The restorative demand should be a class II, III or IV on first or second molars, or premolars. At least two fillings should be from the same tooth group (premolar/molar) in each patient. This will be a split-mouth study, whereby one tooth on one side will be restored using direct technique, and the contra lateral tooth restored using the indirect technique through random allocation. For both direct and indirect restorations, commercially available short-fibre reinforced composite material (Ever X Flow, GC) is used for core material (replacing dentin) and flowable composite material (Gaenial Universal Injectable, GC) for surface (replacing enamel, appr. 2mm thickness from the surface), according the manufacturer´s instructions. Clinical evaluations will be conducted immediately after the final finishing, and after 1 year, 3 years and 5 years. The evaluation will be based on the United States Public Health Service (USPHS) criteria. Descriptive statistics will be used to describe the frequency distributions of the evaluated criteria. To analyse the failure rate for direct vs. indirect restorations, 2x2 tables will be created. Non-parametric statistical procedures will be used due to ordinally structured data for the assessment of the restorations. Mann-Whitney U-test will be used to explore significant differences at different time points between direct and indirect restorations.

DETAILED DESCRIPTION:
Introduction

In dentistry, filling materials are needed repairing damage caused by dental caries as well as for occlusal rehabilitation. Composite restorations can be performed using direct or indirect technique. There are some shortcomings linked with direct technique, such as polymerization shrinkage, and also their manufacturing can be demanding due to circumstances in the oral cavity. Partly due to these, approximately 8 out 10 regular users of dental services need repetitive repair or replacement of old restorations within 5 years. One solution for manufacturing high-qualified and long-lasting restorations is chairside CAD/CAM (computer-aided design and computer-aided manufacturing) technology that includes both subtractive and additive manufacturing techniques. Additive techniques, also called 3D printing techniques, may provide novel possibilities to overcome the challenges linked with the durability of dental fillings. They might be used to fabricate more complex restorations compared to subtractive techniques with a reasonable cost. In 3D printing, successive layers of material are deposited under computer control to create an object layer by layer. The objects, having practically any shape or geometry, are produced from a model or design in an electronic form. The 3D printable models may be created with a CAD software package and in many cases utilize the imaging data by a dental scanner which have become widely available with high resolution. 3D printing may enable higher restoration accuracy compared to subtractive manufacturing techniques, where the accuracy is limited by the milling unit and machining tools. Another benefit is its low material loss. 3D printing process is fast and likely in future to be used chairside at the dental office. Only a few studies addressing the possibilities of 3D printing in dental filling manufacture exist in the current literature. Based on a previous in vitro study by the imvestigators, the accuracy of 3D printing technique is at least at the same level as milling technique in fabrication of dental inlay and onlay fillings, and thus might be a clinically acceptable alternative to the subtractive milling technique. Additional clinical investigations are needed to confirm these findings. The aim of the present study is to compare the success of dental fillings prepared using 3D printing technique to those manufactured with the direct composite technique.

Material and Methods

At total, 100 adult patients are selected from dental care patients of the Health Centre of Kaarina, Kaarina, Finland, as volunteers. Written informed consent forms are obtained from all patients at the beginning of the study. Participation in the study is voluntary and causes no additional costs for the patient.

Each patient requires two Class II, III or IV cavities to be restored in the dentition. The randomizations are performed by noting each tooth to be restored (Fédération Dentaire Internationale [FDI] two-digit code) on one form and the type of restorative system (direct technique vs. indirect technique utilizing 3D printing) on a second. First, a tooth number is drawn blindly. Subsequently, a restorative system is allocated to this tooth by blind drawing. The clinical procedures of cavity preparation and restoration placement are performed by two experienced dentists.

Clinical Evaluation Restorations are rated independently by blinded dentists at the Institute of Dentistry, University of Turku, Finland, who are not involved with the insertion of the indirect and the direct restorations and are unaware of the group status of the fillings. The two evaluators are calibrated against a reference standard. This clinical assessment method results in ordinally structured data for the outcome variables.

Statistical Analysis Power analysis was used to estimate the sample size. In the calculation, the distributions for clinically excellent or acceptable restorations (direct 87% vs. indirect 93%) based on a previous study. Based a previous in vitro study, it was estimated that restorations based on 3D printing technique have at least as high success rate as indirect ceramic restorations, 96%. When the statistical significance was set p <0.05, alpha coefficients 0.05 and beta value 0.2, the sample size n=150 tooth restorations per group was calculated. The number of patients for the study is estimated between 75 (when 4 restorations are performed for each patient) and 150 (2 restorations performed for each patient).

Descriptive statistics are used to describe the frequency distributions of the evaluated criteria. To analyse the failure rate (distributions of Charlie scored versus non-Charlie-scored restorations) for direct vs. indirect restorations, 2x2 tables are created. Non-parametric statistical procedures are used due to ordinally structured data for the assessment of the restorations. Mann-Whitney U-test is used to explore significant differences at different time points between direct and indirect restorations. The same test is used to detect differences between baseline and follow-up registration. The standard value considered to demonstrate statistically significant differences was set at p <0.05.

Ethical issues

Participation in the study is voluntary and requires an informed consent of the patient. The patient has a right to refuse or interrupt his/her participation in the study at any stage. The patients are treated according to the good clinical practices. Quality of the treatment is suspected to be at least at the same level as in normal treatment methods for restorative care. During the study, the patients will have additional check-ups as, which is compensated with economical or other benefits. Patient data are saved in patient registers at the care-providing instances. Research data are saved and analysed anonymously using SPSS 25 (IBM Statistic Viewer) program.

ELIGIBILITY:
Inclusion Criteria:

* presence of cavities, fractures or cosmetic demands
* first or second molars and permanent premolars needing restorations
* at least two class II restorations from the same tooth group (premolar/molar) should be performed in each patient
* the number of restorations of each technique should be equal in each patient

Exclusion Criteria:

* pulp exposure or risk of it during caries removal or cavities with imminent risk of pulp exposure
* spontaneous pain or sensitivity to percussion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The United States Public Health Service (USPHS) criteria; changes during the follow-up period | baseline, and 1 year, 3 years and 5 years after baseline
  The USPHS criteria include the following evaluations: retention, postoperative sensitivity, secondary caries, colour match, anatomical form, marginal discoloration, marginal adaptation, and surface texture. This clinical assessment method results in ordinally structured data for the outcome variables (A, Alpha = excellent result; B, Bravo = acceptable result; C, Charlie = unacceptable, replacement of the restoration necessary).

CONTACTS AND LOCATIONS:
Overall Officials: Kirsi Sipilä, Professor, Study Director — University of Oulu, Finland
Locations (1):
- Research Unit of Oral Health Sciences, University of Oulu, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alharbi N, Wismeijer D, Osman RB. Additive Manufacturing Techniques in Prosthodontics: Where Do We Currently Stand? A Critical Review. Int J Prosthodont. 2017 September/October;30(5):474-484. doi: 10.11607/ijp.5079. Epub 2017 Jul 27. PMID 28750105
- [Background] Ahlholm P, Sipila K, Vallittu P, Jakonen M, Kotiranta U. Digital Versus Conventional Impressions in Fixed Prosthodontics: A Review. J Prosthodont. 2018 Jan;27(1):35-41. doi: 10.1111/jopr.12527. Epub 2016 Aug 2. PMID 27483210
- [Background] Ahlholm P, Sipila K, Vallittu P, Kotiranta U, Lappalainen R. Accuracy of inlay and onlay restorations based on 3D printing or milling technique - a pilot study. Eur J Prosthodont Restor Dent. 2019 May 30;27(2):56-64. doi: 10.1922/EJPRD_01814Ahlholm09. PMID 31046209
- [Background] Astvaldsdottir A, Dagerhamn J, van Dijken JW, Naimi-Akbar A, Sandborgh-Englund G, Tranaeus S, Nilsson M. Longevity of posterior resin composite restorations in adults - A systematic review. J Dent. 2015 Aug;43(8):934-54. doi: 10.1016/j.jdent.2015.05.001. Epub 2015 May 21. PMID 26003655
- [Background] Beuer F, Schweiger J, Edelhoff D. Digital dentistry: an overview of recent developments for CAD/CAM generated restorations. Br Dent J. 2008 May 10;204(9):505-11. doi: 10.1038/sj.bdj.2008.350. PMID 18469768
- [Background] Chochlidakis KM, Papaspyridakos P, Geminiani A, Chen CJ, Feng IJ, Ercoli C. Digital versus conventional impressions for fixed prosthodontics: A systematic review and meta-analysis. J Prosthet Dent. 2016 Aug;116(2):184-190.e12. doi: 10.1016/j.prosdent.2015.12.017. Epub 2016 Mar 2. PMID 26946916
- [Background] Baratieri LN, Canabarro S, Lopes GC, Ritter AV. Effect of resin viscosity and enamel beveling on the clinical performance of Class V composite restorations: three-year results. Oper Dent. 2003 Sep-Oct;28(5):482-7. PMID 14531591
- [Background] Ebert J, Ozkol E, Zeichner A, Uibel K, Weiss O, Koops U, Telle R, Fischer H. Direct inkjet printing of dental prostheses made of zirconia. J Dent Res. 2009 Jul;88(7):673-6. doi: 10.1177/0022034509339988. PMID 19641157
- [Background] Eftekhar Ashtiani R, Nasiri Khanlar L, Mahshid M, Moshaverinia A. Comparison of dimensional accuracy of conventionally and digitally manufactured intracoronal restorations. J Prosthet Dent. 2018 Feb;119(2):233-238. doi: 10.1016/j.prosdent.2017.03.014. Epub 2017 Jun 2. PMID 28578984
- [Background] Garoushi S, Gargoum A, Vallittu PK, Lassila L. Short fiber-reinforced composite restorations: A review of the current literature. J Investig Clin Dent. 2018 Aug;9(3):e12330. doi: 10.1111/jicd.12330. Epub 2018 Feb 25. PMID 29479830
- [Background] Keshvad A, Hooshmand T, Asefzadeh F, Khalilinejad F, Alihemmati M, Van Noort R. Marginal gap, internal fit, and fracture load of leucite-reinforced ceramic inlays fabricated by CEREC inLab and hot-pressed techniques. J Prosthodont. 2011 Oct;20(7):535-40. doi: 10.1111/j.1532-849X.2011.00745.x. Epub 2011 Aug 1. PMID 21806704
- [Background] Lee KY, Cho JW, Chang NY, Chae JM, Kang KH, Kim SC, Cho JH. Accuracy of three-dimensional printing for manufacturing replica teeth. Korean J Orthod. 2015 Sep;45(5):217-25. doi: 10.4041/kjod.2015.45.5.217. Epub 2015 Sep 23. PMID 26445716
- [Background] Leinfelder KF. Evaluation of criteria used for assessing the clinical performance of composite resins in posterior teeth. Quintessence Int. 1987 Aug;18(8):531-6. No abstract available. PMID 3507720
- [Background] Mai HN, Lee KB, Lee DH. Fit of interim crowns fabricated using photopolymer-jetting 3D printing. J Prosthet Dent. 2017 Aug;118(2):208-215. doi: 10.1016/j.prosdent.2016.10.030. Epub 2017 Jan 12. PMID 28089333
- [Background] Mangani F, Marini S, Barabanti N, Preti A, Cerutti A. The success of indirect restorations in posterior teeth: a systematic review of the literature. Minerva Stomatol. 2015 Oct;64(5):231-40. PMID 26094896
- [Background] Nihtila A, Widstrom E, Elonheimo O. Adult heavy and low users of dental services: treatment provided. Swed Dent J. 2016;40(1):21-32. PMID 27464379
- [Background] Opdam NJ, van de Sande FH, Bronkhorst E, Cenci MS, Bottenberg P, Pallesen U, Gaengler P, Lindberg A, Huysmans MC, van Dijken JW. Longevity of posterior composite restorations: a systematic review and meta-analysis. J Dent Res. 2014 Oct;93(10):943-9. doi: 10.1177/0022034514544217. Epub 2014 Jul 21. PMID 25048250
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- Available data/document: Study Protocol — http://www.oulu.fi/medicine/node/52771